CLINICAL TRIAL: NCT03574077
Title: Semi-personalized Smoking Cessation Interventions for Adult Smokers Recruited at Smoking Hotspots: a Pilot Randomized Controlled Trial
Brief Title: Semi-personalized IM Smoking Cessation Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Dr. Man Ping WANG, Assistant Professor, School of Nursing, HKU, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UW15-232
Record Dates: First submitted 2017-11-09; First posted 2018-06-29 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: This pilot randomized controlled trial (RCT) has 2 arms: intervention group A (Group A), and control group (Group B). The participants will be randomly assigned to one of the 2 groups. The investigators will randomly select 12 smoking hotspots (SH) from different locations in Hong Kong Island, Kowloon and New Territories for recruitment (4 in each region). A total of 24 sessions of recruitment activities will be organized to recruit 282 participants. The onsite recruitment and counselling will be conducted by trained SC ambassadors. SC ambassadors will approach smokers using a "foot-in- the-door" technique. Smoking status will be validated using exhaled carbon monoxide (CO) and eligibility will be checked by a short questionnaire.
Who Masked: Outcomes Assessor
Masking Description: All outcome assessors will be blinded to the group allocation, this RCT will be single-blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Instant messaging (Experimental): AWARD advice + NRT sampling + Active referral + Instant Messaging (IM)
  Interventions: Behavioral: Instant Messaging (IM); Behavioral: AWARD advice; Behavioral: NRT sampling; Behavioral: Active referral
- SMS messaging (Active Comparator): AWARD advice + NRT sampling + Active referral + SMS messaging
  Interventions: Behavioral: AWARD advice; Behavioral: NRT sampling; Behavioral: Active referral; Behavioral: SMS messaging

INTERVENTIONS:
Behavioral: Instant Messaging (IM) — Tailored automatic, fix- scheduled regular messages will be sent and counselors will interact with smokers in the intervention group through WhatsApp since initial contact and until 2-month after baseline. The interaction will follow the principle of Motivational Interviewing, which will focus on enabling change through the enhancement of intrinsic motivation and the exploration and resolution of ambivalence. Counsellors will identify discrepancies between participants' thought and their action, support their autonomy, be empathetic towards the participant, avoid confrontation, and adjust to resistance. Any smokers who do not use IM or refuse to receive IM messages will be contacted via SMS messages or telephone calls. For smokers who do not respond to regular messages, 3 additional prompt messages will be sent in the 1st month to initiate a conversation.
  Arms: Instant messaging
Behavioral: AWARD advice — AWARD will be delivered to smokers onsite and this includes: Ask about smoking history, Warn about the high risk, Advise to quit or reduce smoking as soon as possible, Refer smokers to smoking cessation services (with a SC service information card), and Do it again: to repeat the intervention; participants who fail to quit or relapse will be encouraged to quit again (and those who have quit smoking will be encouraged to prevent relapse) during telephone follow-ups. The whole process of AWARD can be delivered within 1 to 2 minutes.
Behavioral: NRT sampling — One-week free nicotine replacement therapy (NRT) sampling (gum or patch) will be disseminated to participants who are interested to try after completing the baseline questionnaire. An NRT use card containing reminders of NRT use and potential side effects will be given. Counselors and research staff will also check the side effects of NRT use during WhatsApp interaction and telephone follow-ups.
Behavioral: Active referral — SC ambassadors will introduce various SC services in Hong Kong (using the SC service information card) and motivate smokers to use the SC services. Written consents will be obtained from smokers who are ready to book the service onsite for transfer of their contact telephone numbers to their chosen service providers. Our research staff will transfer the information to the service providers within a week since the enrollment. For smokers in Group A, our research staff will also assist them to re-book the appointments upon their request at follow-up. SC ambassadors will encourage smokers in Group A who are not ready to book SC service to make an early appointment and assist them at follow-up.
Behavioral: SMS messaging — All smokers will receive fix-schedule general messages on SC through short message service (SMS) since their initial participation until 2-month after baseline. These messages include: (a) brief health warning, (b) benefit of quitting, (c) methods to quit and to cope with craving, and (d) SC services and their effectiveness. General SC messages will be sent twice per week in the 1st month and once per week in the 2nd month after joining this study.
  Arms: SMS messaging

SUMMARY:
Text messaging can provide smokers with quitting methods, information on available smoking cessation (SC) services and social support. This kind of intervention was proven to be effective for smoking cessation. Instant messaging (IM), by sending text and pictures, could provide users with better instantaneous and inexpensive support in their time of need. However, IM intervention is understudied in smoking cessation or other health-related areas to our knowledge, its approaches and efficacy warrant further investigation. This study aims to assess the effect of the combined intervention (nicotine replacement therapy sampling, active referral, and brief advice plus a supportive semi-personalized instant messaging advice) on smoking cessation and to assess the effect of the above interventions on secondary outcomes, including quit intention and attempts, smoking reduction, level of nicotine dependence, use of nicotine replacement therapy (NRT) and SC services.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or above and smoked at least 1 cigarette daily;
2. Hong Kong residents able to read and speak Cantonese;
3. Exhaled carbon monoxide of 4 ppm or above, assessed by a Smokerlyzer;
4. Using a cell phone with instant messaging tool (e.g. WhatsApp, WeChat);
5. Able to use instant messaging tool (e.g. WhatsApp, WeChat) for communication;

Exclusion Criteria:

1. Have psychiatric/ psychological diseases or regular psychotropic medications; and
2. Using SC medication, NRT, other SC services or projects.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Biochemically validated abstinence | 3-month follow-up
  Biochemically validated abstinence (exhaled carbon monoxide <4 ppm and saliva cotinine <= 10 ng/ml)
Biochemically validated abstinence | 6-month follow-up
  Biochemically validated abstinence (exhaled carbon monoxide <4 ppm and saliva cotinine <= 10 ng/ml)

SECONDARY OUTCOMES:
Self-reported 7-day point prevalence abstinence | 3-month and 6-month follow-up
  Self-reported no cigarette smoking (even a single puff) in the past 7 days
Level of nicotine dependence | 3-month and 6-month follow-up
  The Heaviness of Smoking Index, a validated scale, will be used to measure the level of nicotine dependence. This scale consists of 2 questions: (1) how soon after waking up does a participant smoke the first cigarette with responses "within 5 minutes", "6-30 minutes", "31-60 minutes" and "after 60 minutes"; (2) how many cigarettes does a participant smoke in a day with responses "1-10", "11-20" "21-30" and ">30".
Readiness to quit smoking | 3-month and 6-month follow-up
  Readiness to quit smoking will be measured by a question asking the planned quit day based on the Transtheoretical Model with the following responses: within 7days, with 30 days, within 60 days, not yet decided.
Quit attempts | 3-month and 6-month follow-up
  Self-reported quit attempts after enrollment in the study
Smoking reduction | 3-month and 6-month follow-up
  Reduction in the number of cigarettes smoked daily by at least 50% of the baseline amount
NRT use | 3-month and 6-month follow-up
  The amount of nicotine replacement therapy (NRT) used including the sampling received at baseline, NRT received from SC services, NRT bought by participants
SC services used | 3-month and 6-month follow-up
  Smoking cessation service used after enrollment in the study

CONTACTS AND LOCATIONS:
Locations (1):
- School of Nursing, The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Zhao SZ, Wu YS, Chau SL, Fong DYT, Lam TH, Wang MP. Mobile chat-based support plus nicotine replacement therapy sampling to promote smoking cessation for community smokers: A randomized controlled trial. Tob Induc Dis. 2021 Apr 27;19:32. doi: 10.18332/tid/133373. eCollection 2021. PMID 33927586